CLINICAL TRIAL: NCT01034449
Title: Transplantation of Ex-vivo Expanded Human Cord Blood Hematopoietic Stem Cells Expanded: Evaluation of Hematopoietic and Immunologic Reconstitution After a Reduced-intensity Conditioning Regimen
Brief Title: Transplantation of Ex-vivo Expanded Cord Blood Stems Cells
Acronym: GRAPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2008/12
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Malignant Haematological Disease
Keywords: allo graft; cord blood; expansion; reduced-intensity conditioning
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: allogeneic transplant — ex vivo amplification of a unit of placental blood for transplantation

SUMMARY:
This program offers the opportunity to receive an allogeneic transplant to try to control the malignant hematologic in the absence of acceptable conventional donor and with a risk-benefit ratio equivalent to that which would be expected with a transplant from a more conventional donor.

An economy of means in that this method could serve as an alternative to 2 units of placental blood transplantation. The current cost of disposal of a unit of placental blood from a bank is approximately 22000 € (Source: Biomedicine Agency, 2007 rates). The amplification process as controlled by "EFSAL" is 12000 €. Therefore, buying a unit and ex-vivo amplification is more economical. Moreover, the availability of placental blood is not infinite, and the use of one unit per patient will also save resources that can be valuable for certain groups of patients.

In the longer term, methods of amplification of specific immunocompetent cells (from the fraction of CD 34 neg cells) are already being evaluated in the laboratory. They allow to consider a faster recovery, better and more targeted, including cells against the disease for which transplantation is performed.

DETAILED DESCRIPTION:
This is a multicenter prospective non randomized phase 2 clinical trial.

The primary objective is defined by getting a neutrophil count above 500/ml for 3 consecutive days at day 42 after transplantation, in association with complete or partial chimerism on T cells (10 % to 90%).

The secondary objectives are:

* the feasibility of expansion,
* tolerance immediate injection of a graft amplified,
* the payback of a platelet count> 20 000/microlitre without transfusion,
* Incidence of graft loss or rejection within 6 months following transplantation,
* the incidence of acute and chronic GVHD,
* the mortality rate associated with transplantation,
* the incidence of relapse of hematologic malignancies,
* Overall survival,
* Disease-free survival at 1 year post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and < 66 years
* Patient with acute myeloid leukemia (AML) high risk in 1st complete remission:
* CR1 obtained by 2 cycles of chemotherapy,
* unfavorable Cytogenetics
* FLT3 Duplication,
* Or acute myeloid leukemia (AML) in 2nd complete remission,
* Or acute lymphoblastic leukemia (ALL) High-risk 1st complete remission:
* Presence of the translocation t (9; 22),
* Or acute lymphoblastic leukemia (ALL) in 2nd complete remission,
* Or Chronic Myeloid Leukemia (LCM) beyond the 1st chronic phase
* Or Myelodysplasia or with IPSS score with 2 or more
* Or Hodgkin's disease in sensitive relapse or beyond the 2nd complete remission. or following types of lymphoma :
* Diffuse large B lymphoma cells relapsed or refractory after two lines of treatment or after a line with autologous hematopoietic stem cell, or
* Mantle cell lymphoma relapsed or refractory after two lines of treatment or after a line with autologous hematopoietic stem cell
* Others aggressive lymphoma for which an indication of allograft is selected (Burkitt lymphoma, lymphoblastic lymphoma, intravascular lymphoma, ...)
* Lymphoma (low-grade follicular lymphoma, marginal zone lymphoma) in histological transformation.
* Low-grade lymphoma for which an indication of allograft is retained
* Unable to receive myeloablative conditioning because of age (> 45 years) and/or the existence of co-morbidities precluding a myeloablative conditioning (status ECOG > / = 2, DLCO <50%, fungal infection proven or probable in the previous 60 days) and / or prior treatment with total body irradiation at doses above 2 Gy or busulfan doses> 8 mg/kg
* No contra-indication for a transplant in allogeneic non-myeloablative conditioning,
* No HLA-identical sibling,
* Absence of an unrelated donor on national or international registering with a 10/10 allelic matching or a 9/10 allelic matching with the only tolerated mismatches being: HLA-C.
* No unit of placental blood available fulfilling the characteristics of compatibility (HLA compatible at least 4/6 allele or generic) and richness
* Provision of at least 2 units of placental blood, whose compatibility is 4/6, 5/6 or 6/6 and whose richness is before thawing, > 2 x 107 and < 3 to 4 x 107 nucleated cells per/kg.
* Patient affiliated to a social security scheme,
* Free and informed consent signed by the patient and the investigator.

Exclusion Criteria:

* Age <18 and ≥ 66 years
* Malignant myeloid or lymphoid acute or chronic disease without indication for an allogeneic transplant according to the criteria of European Bone Marrow Transplantation Group.
* Able to receive a myeloablative conditioning because of age (<45 years) and the absence of co morbidities (status ECOG> / = 2, DLCO <50%, fungal infection proven or probable in 60 preceding days) and the absence of prior treatment with total body irradiation at doses above 2 Gy or busulfan doses> 8 mg / kg
* Contra indication for a non-myeloablative conditioning,
* HLA-identical sibling available
* Availability of an unrelated donor on a national or international register with 10/10 or 9/10 HLA matching (HLA-C Mismatch tolerated).
* At least one unit of cord blood available with the characteristics of compatibility (HLA compatible at least 4/6 allelic or generic) and richness (before thawing> / = 3 to 4 x 107 nucleated cells/kg recipient, by degree of compatibility)
* Absence of at least 2 units of placental blood, whose compatibility is 4/6, 5/6 / or 6/6 and whose richness before thawing is > 2 x 107 and < 4 x 107 nucleated cells per/kg of recipient.
* Women of childbearing age not using contraception, pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The number of granulocytes, which will be evaluated daily after transplantation. And chimerism to be measured on the cells (total nucleated cells and lymphocytes) from peripheral blood on days 15, 42, 60, 100, 180, 360. | Daily for Blood évaluation and on days 15-42-60-100-180-360 for chimérisme évaluation.

SECONDARY OUTCOMES:
feasibility of expansion | during and after expansion
Immediate tolerance of a graft amplified injection. Determined by measurement of vital parameters during injection of the graft and within 3 hours of observation and clinical tolerance. | during injection of the graft and within 3 hours of observation
The payback of a platelet count> 20 000/microlitre bloodless. Measured by the blood count and platelet daily during hospitalization and at least 2 times a week. | until the payback of the platelet count : measured daily during hospitalization and at least 2 times a week after
The length of hospitalization since the beginning of conditioning until the first exit for more than 2 days. | lenght of hospitalization since the beginning of conditioning
The number of transfusions of red blood cells and platelets during the 1st hospitalization | during the first hospitalization
The incidence of graft loss or rejection within 6 months after transplantation, defined as the installation of a central cytopenia with loss of chimerism | Within 6 months after transplantation
The incidence of acute and chronic GVHD,determined by clinical examination Biopsies of target organs(skin, intestine, liver) will be conducted to confirm the diagnosis if possible. | daily during hospitalization and at least twice weekly until D 100 after transplantation and then weekly or bi-monthly until one year post transplant.
The mortality rate for transplantation in the year following the transplant, | in the year following the transplant
The incidence of relapse of hematologic malignancies, | in the year following the transplant
survival and disease-free survival in the year following the transplant | in the year following the transplant
Monitoring of immune reconstitution. This reconstruction will be followed by determining the rate of immunoglobulin G, M and A and the number of T lymphocytes CD3 +, CD4 + and CD8 + (assessments on days 15, 42, 60, 100, 180, 360). | on days 15, 42, 60, 100, 180, 360

CONTACTS AND LOCATIONS:
Overall Officials: Noel MILPIED, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (3):
- France (3):
  - Service d'hématologie et d'Oncologie Clinique - Hôpital Lapeyronie - 371 avenue du Doyen Gaston GIRAUD, Montpellier
  - Service d'Hématologie, Hôpital Hôtel Dieu, CHU de Nantes - 1 Place Alexis Ricordeau, Nantes
  - Service des maladies du sang - Hôpital Haut-Lévêque - avenue de Magellan, Pessac

REFERENCES:
- [Background] Petersdorf EW. Risk assessment in haematopoietic stem cell transplantation: histocompatibility. Best Pract Res Clin Haematol. 2007 Jun;20(2):155-70. doi: 10.1016/j.beha.2006.09.001. PMID 17448954
- [Background] Koh LP, Chao NJ. Umbilical cord blood transplantation in adults using myeloablative and nonmyeloablative preparative regimens. Biol Blood Marrow Transplant. 2004 Jan;10(1):1-22. doi: 10.1016/j.bbmt.2003.09.009. PMID 14752775
- [Background] Barker JN, Weisdorf DJ, DeFor TE, Blazar BR, McGlave PB, Miller JS, Verfaillie CM, Wagner JE. Transplantation of 2 partially HLA-matched umbilical cord blood units to enhance engraftment in adults with hematologic malignancy. Blood. 2005 Feb 1;105(3):1343-7. doi: 10.1182/blood-2004-07-2717. Epub 2004 Oct 5. PMID 15466923
- [Background] Castello S, Podesta M, Menditto VG, Ibatici A, Pitto A, Figari O, Scarpati D, Magrassi L, Bacigalupo A, Piaggio G, Frassoni F. Intra-bone marrow injection of bone marrow and cord blood cells: an alternative way of transplantation associated with a higher seeding efficiency. Exp Hematol. 2004 Aug;32(8):782-7. doi: 10.1016/j.exphem.2004.05.026. PMID 15308330
- [Background] Shpall EJ, Quinones R, Giller R, Zeng C, Baron AE, Jones RB, Bearman SI, Nieto Y, Freed B, Madinger N, Hogan CJ, Slat-Vasquez V, Russell P, Blunk B, Schissel D, Hild E, Malcolm J, Ward W, McNiece IK. Transplantation of ex vivo expanded cord blood. Biol Blood Marrow Transplant. 2002;8(7):368-76. doi: 10.1053/bbmt.2002.v8.pm12171483.
- [Background] Ljungman P, Urbano-Ispizua A, Cavazzana-Calvo M, Demirer T, Dini G, Einsele H, Gratwohl A, Madrigal A, Niederwieser D, Passweg J, Rocha V, Saccardi R, Schouten H, Schmitz N, Socie G, Sureda A, Apperley J; European Group for Blood and Marrow. Allogeneic and autologous transplantation for haematological diseases, solid tumours and immune disorders: definitions and current practice in Europe. Bone Marrow Transplant. 2006 Mar;37(5):439-49. doi: 10.1038/sj.bmt.1705265. PMID 16444286
- [Background] Brunstein CG, Barker JN, Weisdorf DJ, DeFor TE, Miller JS, Blazar BR, McGlave PB, Wagner JE. Umbilical cord blood transplantation after nonmyeloablative conditioning: impact on transplantation outcomes in 110 adults with hematologic disease. Blood. 2007 Oct 15;110(8):3064-70. doi: 10.1182/blood-2007-04-067215. Epub 2007 Jun 14. PMID 17569820
- [Background] Gluckman E, Rocha V. Donor selection for unrelated cord blood transplants. Curr Opin Immunol. 2006 Oct;18(5):565-70. doi: 10.1016/j.coi.2006.07.014. Epub 2006 Aug 8. PMID 16893632
- [Background] Takahashi S. Leukemia: cord blood for allogeneic stem cell transplantation. Curr Opin Oncol. 2007 Nov;19(6):667-72. doi: 10.1097/CCO.0b013e3282f0e1a1. PMID 17906469
- [Background] Kobari L, Pflumio F, Giarratana M, Li X, Titeux M, Izac B, Leteurtre F, Coulombel L, Douay L. In vitro and in vivo evidence for the long-term multilineage (myeloid, B, NK, and T) reconstitution capacity of ex vivo expanded human CD34(+) cord blood cells. Exp Hematol. 2000 Dec;28(12):1470-80. doi: 10.1016/s0301-472x(00)00557-9. PMID 11146169
- [Background] Duchez P, Dazey B, Douay L, Vezon G, Ivanovic Z. An efficient large-scale thawing procedure for cord blood cells destined for selection and ex vivo expansion of CD34+ cells. J Hematother Stem Cell Res. 2003 Oct;12(5):587-9. doi: 10.1089/152581603322448295. No abstract available. PMID 14594515
- [Background] Dazey B, Duchez P, Letellier C, Vezon G, Ivanovic Z; French Cord Blood Network. Cord blood processing by using a standard manual technique and automated closed system "Sepax" (Kit CS-530). Stem Cells Dev. 2005 Feb;14(1):6-10. doi: 10.1089/scd.2005.14.6. No abstract available. PMID 15725739
- [Background] Ivanovic Z, Duchez P, Dazey B, Hermitte F, Lamrissi-Garcia I, Mazurier F, Praloran V, Reiffers J, Vezon G, Boiron JM. A clinical-scale expansion of mobilized CD 34+ hematopoietic stem and progenitor cells by use of a new serum-free medium. Transfusion. 2006 Jan;46(1):126-31. doi: 10.1111/j.1537-2995.2005.00675.x. PMID 16398741
- [Background] Barker JN, Weisdorf DJ, DeFor TE, Blazar BR, Miller JS, Wagner JE. Rapid and complete donor chimerism in adult recipients of unrelated donor umbilical cord blood transplantation after reduced-intensity conditioning. Blood. 2003 Sep 1;102(5):1915-9. doi: 10.1182/blood-2002-11-3337. Epub 2003 May 8. PMID 12738676
- [Background] Ljungman P, Bregni M, Brune M, Cornelissen J, de Witte T, Dini G, Einsele H, Gaspar HB, Gratwohl A, Passweg J, Peters C, Rocha V, Saccardi R, Schouten H, Sureda A, Tichelli A, Velardi A, Niederwieser D; European Group for Blood and Marrow Transplantation. Allogeneic and autologous transplantation for haematological diseases, solid tumours and immune disorders: current practice in Europe 2009. Bone Marrow Transplant. 2010 Feb;45(2):219-34. doi: 10.1038/bmt.2009.141. Epub 2009 Jul 6. PMID 19584824